CLINICAL TRIAL: NCT01436669
Title: Effectiveness and Feasibility Study of a New Home Full Blood Count Tele-monitoring Device for Cancer Patients Receiving Chemotherapy (ETC1)
Brief Title: Study of Home Full Blood Count (FBC) Telemonitoring Device for Chemotherapy Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Collaborators: The Royal Marsden Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REC 10/H0724/14
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Cancer
Keywords: Chemotherapy use; Home Monitoring
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home Monitoring (Experimental): All participants will receive a home telemonitoring system which will allow cancer patients receiving chemotherapy to test their blood count at home.
  Interventions: Device: Home Telemonitoring System (The Zodiac, Philips Health care)

INTERVENTIONS:
Device: Home Telemonitoring System (The Zodiac, Philips Health care) — Full blood count (FBC) home tele-monitoring system which will allow cancer patients receiving chemotherapy to test their blood count at home (haemoglobin, haematocrit, white cell count and neutrophil count).

SUMMARY:
The Zodiac, a Philips healthcare telemonitoring system has been devised to allow cancer patients receiving chemotherapy to test their blood count at home. It is anticipated that the system will allow patients and clinicians to reduce the toxic effects of chemotherapy by early diagnosis of neutropenia, anaemia and any associated complications of chemotherapy. It is also anticipated that the system will also allow clinicians to better manage the scheduling of chemotherapy regimes.

DETAILED DESCRIPTION:
Philips Healthcare has devised a new home full blood count (FBC) home telemonitoring system which will allow cancer patients receiving chemotherapy to test their blood count at home (haemoglobin, haematocrit, white cell count and neutrophil count). The system will also allow patients to record their temperature and symptoms. The Philips home telemonitoring system is called the Zodiac and consists of a telecommunications hub connected to a haematology analyser. The Hub connects to medical device software running on a remote server which controls the flow of information between the Hub and the clinician. This is designed to enable the patient to self test their full blood count in their home and transmit the data remotely to a clinician for review. In addition to testing their full blood count, the patients can input their temperature and any symptoms they have onto the device. The clinician will then be able to send appropriate instructions back to the patient. The Philips Zodiac system can also send a preprogrammed automated message based on the results of testing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18.
2. Able to give informed written consent in the English language.
3. Diagnosis of cancer and receiving chemotherapy or with a planned chemotherapy start date within 2 weeks of enrolment.
4. Patients who are able to perform finger prick test to obtain capillary blood.

Exclusion Criteria:

1. Inability to give informed consent due to mental capacity or language problems.
2. Patients at risk of bruising or bleeding as a result of their disease or treatment.
3. Patients at risk of bruising or bleeding due to anticoagulants (heparin or warfarin), aspirin or thrombocytopenia (platelet count <80).
4. Patients with diabetes mellitus
5. Patients with peripheral neuropathy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Capillary Blood Sample | 3 times per week for 6 weeks
  To achieve a read out result of a full blood count (haemoglobin, haematocrit, white cell count and neutrophil count) from capillary blood obtained by finger prick and analysed in the Philips Zodiac system that varies by no more than 15% from a sample reported by the standard hospital based laboratory analyser for white cell count, haemoglobin and haematocrit using venous blood.

SECONDARY OUTCOMES:
Number of variances in neutrophil and haemoglobin | 3 times per week for 6 weeks
  To measure the number of variances in the neutrophil and haemoglobin values between the Philips Zodiac system and hospital laboratory analyser, which could result in a different clinical decision being made based on the management of patients at risk of neutropenia and anaemia.
Usability | 3 weeks and 6 weeks of use
  To document the level of satisfaction and feasibility using questionnaires, in the use of the Philips Zodiac system (training, ease of use, performing a blood test and preference for home testing versus hospital testing)
Performance Evaluation | 3 times per week for weeks 1-6
  The questionnaire will assess the patients response to the flow of information via the server software, i.e. the ability of the Philips Zodiac system to provide the patient with a correct automated message or message from a clinician based on the results of the testing; the ability of patients to receive and understand the system messages; and, the satisfaction of patients with the Philips Zodiac System in terms of training issues, ease of use, performing a blood test, performing quality control tests and preference for home testing versus hospital testing.

CONTACTS AND LOCATIONS:
Overall Officials: Nic Kent, Study Director — Philips Healthcare
Locations (1):
- Royal Marsden Hospital, Belmont, Surrey, United Kingdom